CLINICAL TRIAL: NCT04269941
Title: Clinicopathological Characteristics and Prognostic Factors of Gastrointestinal Stromal Tumors Located in the Stomach in Tunisian Patients
Brief Title: Prognostic Factors Affecting Survival of Gastric GIST
Status: Completed | Type: Observational
Sponsor: Université de Sousse (Other)
Responsible Party: Principal Investigator, ammar houssem, Doctor, Université de Sousse
Other Study IDs: U23453
Record Dates: First submitted 2020-02-12; First posted 2020-02-17 (Actual); Last update posted 2020-02-17 (Actual); Status verified 2020-02

CONDITIONS: Gastric GIST

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- prognostic factors of gastrointestinal stromal tumors: for the patient diagnosed with gastic GIST , they underwent subtotal or total gastrectomy.
  Interventions: Other: total or subtotal gastrectomy

INTERVENTIONS:
Other: total or subtotal gastrectomy — resection of the gastric tumor

SUMMARY:
Gastrointestinal stromal tumor (GIST) is the most common non-epithelial mesenchymal tumor of the gastrointestinal tract. Surgical treatment is the only curative therapy for primary localized GIST. This study aimed to identify the clinicopathological characteristics of gastric GISTs and to study the predictive factors for recurrence in Tunisian patients.

DETAILED DESCRIPTION:
The prognosis of gastric GIST depends on various tumor factors with the most important being the mitotic index and tumor necrosis. Imatinib therapy has revolutionized the treatment of advanced GIST.

They have been the subject of much controversy in terms of their histogenesis, classification, treatment and prognosis. GISTs are histologically similar to smooth muscle and nerve tumors such as leiomyomas, leiomyosarcomas or schwannomas. Currently they are well characterized with the recent discovery of the C-KIT gene mutation and the expression by tumor cells of the C-KIT protein.

Moreover, the discovery of this receptor is at the origin of the introduction of a "targeted therapy": an anti-tyrosine kinase molecule having revolutionized the therapeutic management of these tumors. However, the standard curative treatment of GIST remains complete surgical resection with negative margin from the tumor.

ELIGIBILITY:
Inclusion Criteria: patient having gastric GIST

-

Exclusion Criteria:

* patient operated for other gastric tumors

Ages: 10 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: There were 34 patients with the mean age of 58.2 years and male predominance. The disease was localized, locally advanced and metastatic in 26, 6 and 2 cases, respectively. Complete surgical resection was performed in 32 cases.
Sampling Method: Non-Probability Sample
Enrollment: 34 (Actual)
Dates: Start 2000-01-01 (Actual); Primary Completion 2015-01-29 (Actual); Study Completion 2018-01-02 (Actual)

PRIMARY OUTCOMES:
number of patients operated for gastric GIST | 30 days
  the patient having adenocarcinoma or other histopathological type are excluded

CONTACTS AND LOCATIONS:
Overall Officials: ALI BEN ALI, PROFESSOR, Study Director — university of sousse

IPD SHARING:
Plan to Share IPD: Undecided